CLINICAL TRIAL: NCT04833205
Title: Clinical Efficacy and Safety of EGFR-TKI Combined With Nimotuzumab in the Treatment of Leptomeningeal Metastases From Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hui Bu (Other)
Responsible Party: Sponsor-Investigator, Hui Bu, The department of neurology,clincial professor,director, Hebei Medical University
Organization: Hebei Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH005
Record Dates: First submitted 2021-03-01; First posted 2021-04-06 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Leptomeningeal Metastasis; Lung Cancer
Keywords: Leptomeningeal Metastasis; ,Nimotuzumab; Lung Cancer; EGFR-TKI
MeSH Terms: conditions — Meningeal Carcinomatosis; Lung Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leptomeningeal metastases received EGFR-TKI and Nimotuzumab (Experimental): The patients received Nimotuzumab 200 mg,which was diluted in 250mL 0.9% sodium chloride injection, intravenously dripping.And the duration of administration was controlled over 60 min), and the drug was used continuously for 8 weeks.One the other hand,the patient received the third generation of EGFR-TKI
  Interventions: Drug: Nimotuzumab

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab 200 mg was diluted in 250mL 0.9% sodium chloride injection, intravenously dripping, the duration of administration was controlled over 60 min), and the drug was used continuously for 8 weeks
  Other Names: EGFR-TKI

SUMMARY:
Clinical Efficacy and Safety of EGFR-TKI Combined With Nimotuzumab in the Treatment of Leptomeningeal Metastases From Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older, gender not limited;
* A definite diagnosis of Leptomeningeal metastases from lung cancer, including cerebrospinal fluid cytology and/or neuroimaging;
* Have a clear history of lung cancer, including histopathological diagnosis, or cytopathology combined with imaging diagnosis
* Patients who received any of EGFR inhibitors (gefitinib, erlotinib, afatinib, osimertinib etc.) meet the diagnostic criteria for secondary resistance and were in a slow progression stage
* Detection results of cerebrospinal fluid, blood gene or lung tissue specimens showed EGFR mutation, and immunohistochemistry results of cerebrospinal fluid, blood gene or lung tissue showed positive EGFR expression
* Bone marrow, liver, kidneys and blood clotting function are relatively stable

Exclusion Criteria:

* Eastern Cooperative Oncology Group scored > 2 points
* Patients had poor compliance, or for other reasons the investigator considered them unsuitable to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-19 (Estimated); Primary Completion 2022-04-19 (Estimated); Study Completion 2023-04-19 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 2 years
  From the diagnosis of the LM to the time of disease worsen

SECONDARY OUTCOMES:
Overall Survival | 2 years
  From the diagnosis of theLM to the time of death
Incidence of Treatment-Emergent Adverse Events | 8Weeks
  When the Nimotuzumab is used,we will observe if the patients have the allergic reaction,diarrhea ,vomiting and so on.Number of participants with treatment-related adverse events as assessed by CTCAE v4.0"

CONTACTS AND LOCATIONS:
Overall Officials: jiao xue qi, master, Principal Investigator — The Second Hospital of Hebei Medical University
Locations (2):
- China (2):
  - The Second Hospital of Hebei Medical University, Hebei, Shijiazhuang/hebei
  - The Second Hospital of Hebei Medical University, Hebei

IPD SHARING:
Plan to Share IPD: No